CLINICAL TRIAL: NCT01702012
Title: Evaluation of Almased on Glycemic Control and Metabolic Effects in Patients With Type 2 Diabetes
Brief Title: Almased Multi-Center Diabetes Intervention Trial
Acronym: AMDIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of Freiburg (Other); University of Campinas, Brazil (Other); London Metropolitan University (Other); University of Mysore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00020672
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Diabetes-Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almased Meal Replacement Powder (Experimental): Participants assigned to this arm will receive the Almased meal replacement powder and will be asked to replace one meal per day during the first 6 months of participation. During the second 6 months, participants will be allowed to choose whether to continue using the product to replace a meal or to use the product as a supplement prior to meals.
  Interventions: Dietary Supplement: Almased Meal Replacement Powder
- Lifestyle Intervention (Active Comparator): Participants randomized to this group will receive 5 group sessions in the first two months of participation and 5 additional group sessions in the last two months. These group sessions will focus on lifestyle behavior changes for weight loss and management including goal-setting, calorie balance, general nutrition, and physical activity.
  Interventions: Behavioral: Group-Based Lifestyle Intervention

INTERVENTIONS:
Dietary Supplement: Almased Meal Replacement Powder — Commercially available meal replacement product that contains soy protein, honey, yogurt, and amino acids. Participants assigned to this arm will receive the Almased meal replacement product and will be asked to replace one meal per day during the first 6 month. During the second 6 months, they will be allowed to choose to continue using the Almased as a meal replacement or to use it as a supplement prior to meals.
  Arms: Almased Meal Replacement Powder
Behavioral: Group-Based Lifestyle Intervention
  Arms: Lifestyle Intervention

SUMMARY:
A 12 month multi-center randomization controlled study. Participants will be randomized to either a lifestyle education program or a meal replacement regimen with Almased, after an initial examination of eligibility criteria.

Primary outcome-HbA1c

DETAILED DESCRIPTION:
Age 21 + Male/Female gender Type 2 Diabetes Non-insulin dependent BMI 25-40 kg/m HbA1c 7.5-10%

ELIGIBILITY:
Inclusion Criteria:• Gender: Men and women are eligible

* Type 2 diabetes mellitus: Diabetes mellitus will be determined by medical records, current treatment, verification from personal health care provider, or test results meeting the 2010 American Diabetes Association criteria of fasting glucose ≥126 mg/dl, symptoms of hyperglycemia with casual plasma glucose > 200 mg/dl or two-hour plasma glucose ≥200 mg/dl after a 75 gram oral glucose load. Individuals who have a clinical history strongly suggestive of type 1 diabetes will be excluded. Individuals taking oral hypoglycemic medication with diet and exercise are eligible. Subjects taking insulin will not be eligible for entry into the study.
* Body mass index: Overweight and obese individuals, with body mass index 25 - 40 kg/m2, are eligible. Weight loss is recommended for overweight diabetic participants with one or more cardiovascular risk factors.
* Age: Individuals older than 21 years are eligible.
* Ethnicity: All ethnic groups are eligible for the study.
* Blood pressure: AMDIT will enroll individuals whose blood pressure is under at least moderate control. For safety purposes, moderate control will be defined in this study as systolic values under 160 mm/Hg and diastolic values under 100 mm/Hg. Individuals whose blood pressure exceeds these levels during screening will be advised to seek treatment and may be re-evaluated following initiation of antihypertensive treatment.
* Glycemic control: AMDIT will enroll individuals whose HbA1c is between 7.5 and 10%. Individuals whose HbA1c exceeds this level may require more urgent care and will be told to seek treatment and may also be re-evaluated for inclusion.
* Lipid control: Individuals with a fasting triglycerides concentration less than 500 mg/dl are eligible.
* Willingness to participate: Participants must be willing to be randomized to either Almased or the Lifestyle Intervention and to follow the protocol to which they have been assigned. Individuals must be willing to modify their diet and their activity if they are assigned to the Lifestyle Intervention.

Exclusion Criteria:• Unable or unwilling to give informed consent or communicate with local study staff;

* Psychotic disorders or bipolar disorders, hospitalization for depression in past six months;
* Self-report of alcohol or substance abuse within the past twelve months, current consumption of more than 14 alcoholic drinks per week, and/or current acute treatment or rehabilitation program for these problems;
* Plans to relocate to an area not served by AMDIT or travel plans that do not permit full participation in the study;
* Known allergies to soy or dairy;
* Current use of medications for weight loss;
* Self-reported inability to walk two blocks;
* History of bariatric surgery, small bowel resection, or extensive bowel resection;
* Chronic treatment with systemic corticosteroids as weight gain associated with steroids may interfere with the intervention goals;
* Candidates who have definite plans to move out of the area within the study period;
* Candidates with any dietary practice, behavior, or attitude that would substantially limit adherence to the intervention;
* Currently pregnant or nursing;
* Cancer requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis (e.g. Stage 1 cervical cancer);
* HIV positive (self-report), due to effects on weight and body composition of HIV and medications used to treat HIV;
* Active tuberculosis (self-report);
* Cardiovascular or cardiopulmonary disease including a heart attack or procedure within the past three months; participation in a cardiac rehabilitation program within last three months; stroke or history/treatment for transient ischemic attacks in the past three months; documented history of pulmonary embolus in past six months; unstable angina pectoris or angina pectoris at rest; known history of cardiac arrest; known history of complex ventricular arrhythmia at rest or with exercise; known history of uncontrolled atrial fibrillation (heart rate of 100 beats per minute or more); known history of NYHA Class III or IV congestive heart failure; known history of acute myocarditis, pericarditis or hypertrophic myocardiopathy; known history of clinically significant aortic stenosis; known history of left bundle branch block or cardiac pacemaker unless evaluated by a cardiologist; cardiac defibrillator; heart transplant; known history of aortic aneurysm of at least 7 cm in diameter or aortic aneurysm repair;
* Renal disease: urine dipstick protein of 4+ (equivalent to approximately > 1 g/day), serum creatinine exceeding 1.4 mg/dl (women) or 1.5 mg/dl (men), or currently receiving dialysis;
* Known history of chronic obstructive pulmonary disease that would limit ability to follow the protocol;
* Self-reported chronic hepatitis B or C or cirrhosis;
* Inflammatory bowel disease requiring treatment in the past year;
* Known history of Cushing's syndrome (clinic diagnosis or self-report);
* Known history of Acromegaly (clinical diagnosis or self-report);
* Amputation of lower limbs as result of non-traumatic causes;
* Any major organ transplant (does not include cornea or hair transplants);
* Conditions not specifically mentioned above may serve as criteria for exclusion at the discretion of the clinical site.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (%) | 2, 4, 6, 8, 10, and 12 months

SECONDARY OUTCOMES:
Change in HOMA IR Index | 2, 4, 6, 8, 10, and 12 months
  measure changes in Homeostasis Model of Insulin Resistance
Change in fasting blood glucose (mg/dl) | 2, 4, 6, 8, 10, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mara Z Vitolins, DrPH MPH RD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No